CLINICAL TRIAL: NCT01083628
Title: Automated Text Messaging to Increase Engagement in Cognitive Behavioral Therapy (CBT) for Depression
Brief Title: Text Messaging and Cognitive Behavioral Therapy for Depression
Acronym: HealthySMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 68556-35551-01
Record Dates: First submitted 2010-02-19; First posted 2010-03-10 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Depression
Keywords: mhealth; depression; latinos; text messaging; CBT; SMS
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group CBT for Depression with MoodText' (Experimental): Group cognitive behavioral therapy utilizing the BRIGHT manual for depression along with automated text messaging for mood monitoring and reminder of session content
  Interventions: Behavioral: Group CBT for Depression with MoodText
- Group CBT for Depression (Active Comparator): Standard group cognitive behavioral therapy utilizing the BRIGHT manual for depression
  Interventions: Behavioral: Group CBT for Depression

INTERVENTIONS:
Behavioral: Group CBT for Depression with MoodText — Mobile phone based text messaging to inquire about mood, cognitions, and behaviors on a daily basis.
  Other Names: Group CBT for Depression with HealthySMS
  Arms: Group CBT for Depression with MoodText'
Behavioral: Group CBT for Depression — Standard group CBT for depression using BRIGHT manual
  Arms: Group CBT for Depression

SUMMARY:
This study aims to asses whether adding automated text messaging to group cognitive behavioral therapy for depression increases engagement which may lead to improved outcomes.

DETAILED DESCRIPTION:
Background: Cognitive Behavioral Therapy (CBT) for depression is efficacious, but effectiveness is limited when implemented in low-income settings due to engagement difficulties including nonadherence with skill-building homework and early discontinuation of treatment. Automated messaging can be used in clinical settings to increase dosage of depression treatment and encourage sustained engagement with psychotherapy.

Objectives: The aim of this study was to test whether a text messaging adjunct (mood monitoring text messages, treatment-related text messages, and a clinician dashboard to display patient data) increases engagement and improves clinical outcomes in a group CBT treatment for depression. Specifically, the investigators aim to assess whether the text messaging adjunct led to an increase in group therapy sessions attended, an increase in duration of therapy attended, and reductions in Patient Health Questionnaire-9 item (PHQ-9) symptoms compared with the control condition of standard group CBT in a sample of low-income Spanish speaking Latino patients.

Methods: Patients in an outpatient behavioral health clinic were assigned to standard group CBT for depression (control condition; n=40) or the same treatment with the addition of a text messaging adjunct (n=45). The adjunct consisted of a daily mood monitoring message, a daily message reiterating the theme of that week's content, and medication and appointment reminders. Mood data and qualitative responses were sent to a Web-based platform (HealthySMS) for review by the therapist and displayed in session as a tool for teaching CBT skills.

ELIGIBILITY:
Inclusion Criteria:

* Participation in CBT group at San Francisco General Hospital

Exclusion Criteria:

* Active suicidality
* Active and severe psychosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Aguilera, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aguilera A, Berridge C. Qualitative feedback from a text messaging intervention for depression: benefits, drawbacks, and cultural differences. JMIR Mhealth Uhealth. 2014 Nov 5;2(4):e46. doi: 10.2196/mhealth.3660. PMID 25373390

RESULTS

PARTICIPANT FLOW:
Groups:
- Group CBT With Text Messaging Adjunct: Group CBT for Depression with MoodText: Mobile phone based text messaging to inquire about mood, cognitions, and behaviors on a daily basis.
Period: Overall Study
Arm/Group | Group CBT With Text Messaging Adjunct | Group CBT for Depression
Started | 45 | 40
Completed | 45 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group CBT With Text Messaging Adjunct | Group CBT for Depression | Total
Number analyzed (Participants) | 45 | 40 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 40 | 85
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.71 (11.55) | 51.83 (11.73) | 51.75 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 29 | 67
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 40 | 85
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 40 | 85
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 (Patient Health Questionnaire - 9) is commonly used to screen for depression and to monitor progression of depressive symptoms over time. The scores represent the following depression severity: 0-4: minimal depression, 5-9: mild depression, 10-14: moderate depression, 15-19: moderately severe, 20-27: severe. A score of 10 is often recommended as the cut-off score for diagnosing an episode of depression that may require treatment.
  units on a scale | 13.36 (5.96) | 13.13 (4.99) | 13.25 (5.68)

OUTCOME MEASURES:

1. Primary Outcome: PHQ-9 Depression Symptoms
Description: The PHQ-9 (Patient Health Questionnaire - 9) is commonly used to screen for depression and to monitor progression of depressive symptoms over time. The scores represent the following depression severity: 0-4: minimal depression, 5-9: mild depression, 10-14: moderate depression, 15-19: moderately severe, 20-27: severe. A score of 10 is often recommended as the cut-off score for diagnosing an episode of depression that may require treatment.
Time Frame: 16 weeks
Population: The number of participants analyzed in this intention-to-treat analyses represents the number of participants that provided PHQ-9 scores at the end of the study period, at 16 weeks. Because the PHQ-9 was filled in during psychotherapy sessions, this number is smaller than the original sample (n=44, n=38) due to patient drop-out of psychotherapy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group CBT With Text Messaging Adjunct | Group CBT for Depression
Number analyzed (Participants) | 18 | 9
units on a scale | 6 (4.2) | 12.67 (6.4)

2. Secondary Outcome: Attendance
Description: Number of sessions attended
Time Frame: 16 weeks
Population: For the attendance analyses, 3 patients (1 in the intervention and 2 in the control) were excluded, because the study ended before these patients had been offered 16 sessions of psychotherapy.
Measure: Median (Standard Deviation); unit: sessions
Arm/Group | Group CBT With Text Messaging Adjunct | Group CBT for Depression
Number analyzed (Participants) | 44 | 38
sessions | 6 (2.3) | 2.5 (1.4)

3. Secondary Outcome: Duration of Therapy Attended
Description: Number of weeks until patients dropped out of therapy
Time Frame: 16 weeks
Population: For the duration of therapy analyses, 3 patients (1 in the intervention and 2 in the control) were excluded, because the study ended before these patients had been offered 16 sessions of psychotherapy.
Measure: Median (Full Range); unit: weeks
Arm/Group | Group CBT With Text Messaging Adjunct | Group CBT for Depression
Number analyzed (Participants) | 44 | 38
weeks | 13.5 [1 to 16] | 3 [1 to 16]

ADVERSE EVENTS:
Arm/Group | Group CBT With Text Messaging Adjunct | Group CBT for Depression
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/40
Other Adverse Events (participants affected / at risk) | 0/45 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No